CLINICAL TRIAL: NCT00806182
Title: Cytokines as Biomarkers and Therapeutic Targets in Paraneoplastic Opsoclonus-Myoclonus Syndrome (OMS)
Brief Title: Study of Cytokines in Children With Opsoclonus-Myoclonus Syndrome
Acronym: OMS
Status: Completed | Type: Observational
Sponsor: National Pediatric Neuroinflammation Organization, Inc. (Other)
Responsible Party: Principal Investigator, Michael R. Pranzatelli, M.D., Director, National Pediatric Neuroinflammation Organization, Inc.
Other Study IDs: Thrasher Award 02826-2
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Opsoclonus-myoclonus Syndrome
Keywords: paraneoplastic; neuroblastoma; Kinsbourne syndrome; autoimmune disease; immunotherapy; ataxia
MeSH Terms: conditions — Opsoclonus-Myoclonus Syndrome; Neuroblastoma; Autoimmune Diseases; Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum, plasma, cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric case-controls: These are children who underwent lumbar puncture and blood drawing for diagnostic testing for non-inflammatory neurological or non-neurological disorders, and whose samples were retrieved from the clinical lab under a linked Institutional Review Board (IRB) protocol.
- Pediatric OMS: These are patients treated by the P.I. based on clinical decision making, not a clinical trial (this is an observational study). The types of treatments are varied, and, on the initial evaluation, the patients may be untreated or already tried on various immunotherapies. They range from monotherapy with steroids, ACTH, or IVIg, to disease modifying agents, such as rituximab, cyclophosphamide, and other chemotherapy, typically adjunctively or as combination therapy.

SUMMARY:
The purpose of this study is to determine if cytokines, inflammatory mediators, are increased in spinal fluid and blood, correlate with disease activity, and could serve as biomarkers or therapeutic targets in children with opsoclonus-myoclonus syndrome (OMS), an autoimmune complication of the tumor neuroblastoma.

DETAILED DESCRIPTION:
In this translational research, immunological mechanisms that underlie the assault of the immune system on the brain in paraneoplastic opsoclonus-myoclonus syndrome (OMS) are under evaluation. To test our principal hypothesis that there is an imbalance of pro-inflammatory (Th1) and anti-inflammatory (Th2) cytokines in OMS, a comprehensive cytokine panel will be measured by enzyme-linked immunosorbent assay (ELISA) and multiplexed fluorescent bead-based immunoassay detection (LUMINEX 100 Lab MAP system)in blood and cerebrospinal fluid (CSF) of 400 children. To test the second hypothesis that cytokines could serve as biomarkers of disease activity in OMS, cytokine concentrations will be correlated with clinical variables, such as disease severity, OMS duration, prior relapses, and remissions, as well as immunological variables, such as lymphocyte subset analysis. The cytokine 'biomarker profile' could aid decision making for early intervention by identifying children at high risk for relapse and poor outcome and allow targeting of the most implicated inflammatory cytokines by cytokine therapies. To test our third hypothesis that lack of response to immunotherapy is due in part to failure to increase the expression of anti-inflammatory Th2 cytokines, we will make paired pre/post comparisons of the impact of immunotherapies given in the course of clinical care [steroids, adrenocorticotropin (ACTH), intravenous immunoglobulins (IVIg), rituximab, chemotherapy, other drugs, combinations] on the cytokine and clinical profile. This research could lead to the application of commercially-available cytokines and cytokine blockers or to the development of new ones for OMS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OMS

Exclusion Criteria:

* Equivocal diagnosis
* Contraindications to lumbar puncture
* Treatment with agents outside the scope of the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Referrals to National Pediatric Myoclonus Center Website, www.omsusa.org
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Reduction in inflammatory cytokines | 6 and 12 months
  Reduction in the concentration of inflammatory chemokines/cytokines between clinical time points

SECONDARY OUTCOMES:
Correlation of cytokine concentration and clinical severity score. | 6 and 12 months
  Statistical correlation of chemokine/cytokine concentration with OMS motor severity as measured using the OMS video evaluation scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Pranzatelli, MD, Principal Investigator — National Pediatric Neuroinflammation Organization, Inc.; Elizabeth D Tate, FNP, MN, Study Director — National Pediatric Neuroinflammation Organization, Inc.
Locations (1):
- National Pediatric Myoclonus Center, Formerly at Dept. of Neurology, Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pranzatelli MR, Tate ED, Hoefgen ER, Swan JA, Colliver JA. Therapeutic down-regulation of central and peripheral B-cell-activating factor (BAFF) production in pediatric opsoclonus-myoclonus syndrome. Cytokine. 2008 Oct;44(1):26-32. doi: 10.1016/j.cyto.2008.06.001. Epub 2008 Aug 9. PMID 18675552
- [Background] Pranzatelli MR, Travelstead AL, Tate ED, Allison TJ, Moticka EJ, Franz DN, Nigro MA, Parke JT, Stumpf DA, Verhulst SJ. B- and T-cell markers in opsoclonus-myoclonus syndrome: immunophenotyping of CSF lymphocytes. Neurology. 2004 May 11;62(9):1526-32. doi: 10.1212/wnl.62.9.1526. PMID 15136676
- [Result] Pranzatelli MR, Tate ED, McGee NR, Colliver JA. Cytokines, cytokine antagonists, and soluble adhesion molecules in pediatric OMS and other neuroinflammatory disorders. J Neurol Sci. 2013 Mar 15;326(1-2):53-8. doi: 10.1016/j.jns.2013.01.011. Epub 2013 Feb 4. PMID 23380454
- [Result] Pranzatelli MR, Tate ED, McGee NR, Travelstead AL, Verhulst SJ, Ransohoff RM. Expression of CXCR3 and its ligands CXCL9, -10 and -11 in paediatric opsoclonus-myoclonus syndrome. Clin Exp Immunol. 2013 Jun;172(3):427-36. doi: 10.1111/cei.12065. PMID 23600831
- [Result] Pranzatelli MR, Tate ED, McGee NR, Colliver JA. Pediatric reference ranges for proinflammatory and anti-inflammatory cytokines in cerebrospinal fluid and serum by multiplexed immunoassay. J Interferon Cytokine Res. 2013 Sep;33(9):523-8. doi: 10.1089/jir.2012.0132. Epub 2013 May 9. PMID 23659672
- [Result] Pranzatelli MR, Tate ED, McGee NR, Ransohoff RM. CCR7 signaling in pediatric opsoclonus-myoclonus: upregulated serum CCL21 expression is steroid-responsive. Cytokine. 2013 Oct;64(1):331-6. doi: 10.1016/j.cyto.2013.05.020. Epub 2013 Jun 10. PMID 23764550
- [Result] Pranzatelli MR, Tate ED, McGee NR, Verhulst SJ. CSF neurofilament light chain is elevated in OMS (decreasing with immunotherapy) and other pediatric neuroinflammatory disorders. J Neuroimmunol. 2014 Jan 15;266(1-2):75-81. doi: 10.1016/j.jneuroim.2013.11.004. Epub 2013 Nov 16. PMID 24342231
- [Result] Pranzatelli MR, Tate ED, Travelstead AL, Verhulst SJ. Chemokine/cytokine profiling after rituximab: reciprocal expression of BCA-1/CXCL13 and BAFF in childhood OMS. Cytokine. 2011 Mar;53(3):384-9. doi: 10.1016/j.cyto.2010.12.004. Epub 2011 Jan 5. PMID 21211990
- [Result] Pranzatelli MR, Tate ED, McGee NR, Colliver JA, Ransohoff RM. CCR4 agonists CCL22 and CCL17 are elevated in pediatric OMS sera: rapid and selective down-regulation of CCL22 by ACTH or corticosteroids. J Clin Immunol. 2013 May;33(4):817-25. doi: 10.1007/s10875-013-9867-4. Epub 2013 Jan 23. PMID 23340773
- [Result] Pranzatelli MR, Tate ED, McGee NR, Travelstead AL, Colliver JA, Ness JM, Ransohoff RM. BAFF/APRIL system in pediatric OMS: relation to severity, neuroinflammation, and immunotherapy. J Neuroinflammation. 2013 Jan 16;10:10. doi: 10.1186/1742-2094-10-10. PMID 23324534
- [Result] Pranzatelli MR, Tate ED, McGee NR, Travelstead AL, Ransohoff RM, Ness JM, Colliver JA. Key role of CXCL13/CXCR5 axis for cerebrospinal fluid B cell recruitment in pediatric OMS. J Neuroimmunol. 2012 Feb 29;243(1-2):81-8. doi: 10.1016/j.jneuroim.2011.12.014. Epub 2012 Jan 20. PMID 22264765